CLINICAL TRIAL: NCT02575859
Title: Pilot Study of Adjuvant Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Patients With Colorectal Cancer at High Risk for the Development of Metachronous Peritoneal Metastases
Brief Title: Adjuvant HIPEC to Prevent Colorectal Peritoneal Metastases in High-risk Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 35/13
Record Dates: First submitted 2015-09-21; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Neoplasm; Metastasis
Keywords: HIPEC; peritoneal lavage
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Cisplatin; Mitomycin; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjuvant HIPEC (Experimental): Adjuvant HIPEC will be performed simultaneously with primary tumor resection in patients undergoing curative surgery for primary colorectal cancer associated with risk factors for the development of metachronous peritoneal metastases.
  Interventions: Drug: adjuvant HIPEC; Procedure: surgery
- Matched control (No Intervention): Comparable controls will be retrospectively selected from patients undergoing curative surgery for colorectal cancer at the National Cancer Institute (Milan, Italy) during the same period.
  Every single control patient will be matched with a.patient in HIPEC group according to the following criteria: i) risk-factor for metachronous PM (minimal synchronous PM vs. ovarian metastases vs. pathological tumor [pT] stage (pT4a/b); ii) pathological node (pN) stage (pN0 vs. pN1/2); iii) grading (well/moderately vs. poorly differentiated); iv) histological subtype (adenocarcinoma vs. mucinous/signet ring cell carcinoma); v) sex; vi) age (+/-5 years). The investigators will be blinded to patient outcomes during the process.

INTERVENTIONS:
Drug: adjuvant HIPEC — Closed-abdomen HIPEC with cisplatin (25 mg/m2/l of perfusate) and mitomycin-C (3•3 mg/m2/l of perfusate) at 42•5°C for 60 minutes. Perfusate volume: 4-6 l.
  Other Names: Cisplatin, mitomycin-C
  Arms: Adjuvant HIPEC
Procedure: surgery — Colon resections for primary tumors were performed according to the oncologic principles of adequate lymph-adenectomy. Complete adhesiolysis, resection of falciform hepatic ligament, greater and lesser omentectomy were performed in all patients to ensure optimal perfusion during the HIPEC. Tumor deposits on visceral and parietal surfaces were surgically removed by formal peritonectomy procedures and/or organ resections, as needed.
  Arms: Adjuvant HIPEC

SUMMARY:
The prognosis of peritoneal metastases from colorectal cancer has recently improved with cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (HIPEC). Although outcomes are further improved when early stage peritoneal metastases are treated, adjuvant HIPEC has not yet been thoroughly addressed. This prospective pilot study assessed feasibility, safety and efficacy of HIPEC performed simultaneously with primary curative surgery in colorectal cancer patients with primary tumor-related risk-factors for the development of metachronous peritoneal metastases.

DETAILED DESCRIPTION:
BACKGROUND Peritoneal surfaces are the second most common site of disease progression for colorectal cancer (CRC), following liver metastases. Historically, prognosis of CRC peritoneal metastases (PM) was only about 6 months with palliative systemic chemotherapy or supportive care. Survival improvements have been reported with cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (CRS/HIPEC). However, CRS/HIPEC is more effective and safe when early-stage CRC-PM are treated and most patients are not suitable for CRS/HIPEC, due to extensive peritoneal and/or systemic disease. Also, in the palliative setting, modern systemic therapies appear to be less effective for PM, than non-PM metastatic CRC and absence of symptoms and current limitations of imaging hamper early diagnosis and treatment of PM. These points would support the use of adjuvant HIPEC to prevent the outgrowth of occult peritoneal seeding into macroscopic disease.

STUDY DESIGN This tudy to assesses feasibility and safety of an integrated approach of curative surgery and adjuvant HIPEC performed at the same time as primary surgery in patients with primary CRC at high risk for the development of metachronous PM. Patients are prospectively selected on the base of preoperative clinical and radiological work-up. At surgery, careful exploration of all peritoneal the cavity, and intra-operative pathological examination are carried out to confirm clinical-pathological risk-factors for PM development Standard adjuvant systemic chemotherapy is intended in the postoperative setting. A matched control group will be selected among patients with colorectal cancer undergoing curative surgery and standard adjuvant systemic chemotherapy at the same institution and during the same period.

STUDY POPULATION Patients with colorectal cancer undergoing intentionally curative resection for primary tumors infiltrating the visceral serosa (T4a) or directly invading adjacent organs (T4b), with positive peritoneal washing cytology or resected ovarian or minimal peritoneal metastases.

INTERVENTION Adjuvant HIPEC procedure is performed under general anaesthesia after the completion of the surgical procedures. Colon resections for primary tumors are performed according to the oncologic principles of adequate lymph-adenectomy.Greater and lesser omentectomy and adhesiolysis (if necessary) are performed routinely to ensure optimal perfusion during the HIPEC. Tumor deposits on visceral and parietal surfaces are surgically removed by formal peritonectomy procedures and/or organ resections, as needed. HIPEC is performed with cisplatin (25 mg/m2/l of perfusate) and mitomycin-C (3•3 mg/m2/l of perfusate) at 42•5°C for 60 minutes according to the closed-abdomen .technique.

OUTCOMES Primary end-point is the sensitivity and false positive rate of preoperative/intraoperative assessment of primary tumor-related risk-factors for the development of peritoneal metastases in patients with colorectal cancer undergoing curative surgery..Secondary endpoints are number of participants with adverse events as a measure of safety and tolerability, Cumulative incidence of PM, overall and progression-free survival are assessed in comparison with matched controls.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed colorectal carcinoma;
* curative surgery;
* presence of at least one of the following risk-factors for the development of metachronous PM:

  * minimal synchronous PM (nodules ≤1cm in the omentum and/or close to the primary tumor), completely resected at the same time as primary tumor;
  * synchronous ovarian metastases, also resected at the same time as primary tumor;
  * primary tumor either penetrating visceral peritoneum (T4a),
  * primary tumor directly invading other organs (T4b);
* signature of an informed consent form.
* intention to start adjuvant systemic therapy and postoperative follow-up;
* performance status ≤2 according to the Eastern Cooperative Oncology Group score;
* no significant co-morbidities.
* no active sepsis
* no impaired cardiac function (history of previous cardiac failure, or ejection fraction <40%)
* no impaired renal function (serum creatinin > 1.5 normal value or creatinin clearance < 60 mL/min);
* no impaired hepatic function (serum glutamic oxaloacetic transaminase, serum glutamic pyruvic transaminase, bilirubin > 1.5 normal value);
* no impaired bone marrow function (leucocytes < 4000/mm3 ; neutrophils < 1500/mm3; platelet < 80000/mm3)
* no impaired lung function (diagnosis of severe chronic obstructive pulmonary disease , or forced expiratory volume at one second < 50% or a diffusion capacity of lung for carbon monoxide < 40% age adjusted).

Exclusion Criteria:

* extensive PM (nodules >1cm, and/or nodules outside the omentum and/or beyond the close vicinity of the primary tumor);
* extra-abdominal/hepatic metastases;
* emergency presentation (bleeding, perforated, or occlusive primary);
* bleeding diathesis or coagulopathy
* history of previous neoplasm during the past three years, excluding skin spinocellular/basocellular carcinoma;
* preoperative pelvic radio-chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2010-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Positive predictive value of preoperative/intraoperative assessment of primary tumor-related risk factors for the development of metachronous peritoneal metastases in patients undergoing curative surgery for colorectal cancer. | The primary outcome measure is assessed at an average of one week after the operation, at the time the pathological examination of surgical specimens is expected to be completed.
  The presence versus absence of primary tumor-related risk-factors for the development of metachronous peritoneal metastases, as assessed during the preoperative/intraoperative phase, is compared with the findings of the pathological examination of surgical specimens.

SECONDARY OUTCOMES:
Number of patients with postoperative treatment-related adverse events. | 60 days
  All-type adverse events occurring within 60 days from surgery and adjuvant HIPEC (including surgical complications and systemic toxicities) will be recorded and graded according to the Common Terminology Criteria for Adverse Events of the National Institute of Health (version 4.0).
Peritoneal progression-free survival | 36 months
  Peritoneal progression-free survival is calculated from the day of surgery and HIPEC to the date of death for any cause, or first recurrence involving the peritoneum..

OTHER OUTCOMES:
Overall survival | 36 months
  Overall survival is dated from the day of surgery with HIPEC to the time of death for any cause.
Progression-free survival | 36 months
  Progression-free survival is dated from the day of surgery with HIPEC to the time of postoperative disease progression involving any site, including peritoneal surfaces

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Deraco, MD, Study Director — Fondazione IRCCS Istituto Nazionale Tumori, Milano

REFERENCES:
- [Result] Virzi S, Iusco D, Baratti D, Bonomi S, Grassi A, Kusamura S, Deraco M. Pilot study of adjuvant hyperthermic intraperitoneal chemotherapy in patients with colorectal cancer at high risk for the development of peritoneal metastases. Tumori. 2013 Sep-Oct;99(5):589-95. doi: 10.1177/030089161309900505. PMID 24362862
- [Derived] Baratti D, Kusamura S, Iusco D, Gimondi S, Pietrantonio F, Milione M, Guaglio M, Bonomi S, Grassi A, Virzi S, Leo E, Deraco M. Hyperthermic Intraperitoneal Chemotherapy (HIPEC) at the Time of Primary Curative Surgery in Patients with Colorectal Cancer at High Risk for Metachronous Peritoneal Metastases. Ann Surg Oncol. 2017 Jan;24(1):167-175. doi: 10.1245/s10434-016-5488-5. Epub 2016 Aug 12. PMID 27519353